CLINICAL TRIAL: NCT06417489
Title: Evaluation of Efficacy and Safety of Combination Therapy of Henagliflozin Proline, Retagliptin and Metformin Compared to Sequential Metformin Therapy in Newly Diagnosed Type 2 Diabetes Patients
Brief Title: Evaluation of Efficacy and Safety of Combination Therapy of Henagliflozin Proline, Retagliptin and Metformin in New Diagnosed Type 2 Diabetes Patients
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2024-165-002
Record Dates: First submitted 2024-05-11; First posted 2024-05-16 (Actual); Last update posted 2024-05-16 (Actual); Status verified 2024-05

CONDITIONS: Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Combined Modality Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Combination therapy (Experimental): Henagliflozin Proline 10 mg qd+Regagliptin 100 mg qd+Metformin 500mg bid. The dose of metformin from the first to second week is 500mg bid, and the dose from the third to fourth week is 1000mg bid. If the maximum dose of metformin cannot be tolerated, the researcher shall increase the dosage according to the patient's tolerance situation. The minimum dose is 1000mg/day.
  Interventions: Drug: Combination therapy
- Sequential treatment group (Active Comparator): Metformin, the dose from the first to second week is 500mg bid, and the dose from the third to fourth week is 1000mg bid. If the maximum dose of metformin cannot be tolerated, the researcher shall increase the dosage according to the patient's tolerance situation. The minimum dose is 1000mg/day. After the fourth week of treatment, blood glucose levels were measured. For those whose blood glucose levels did not meet the standard (fasting blood glucose (FPG)>7mmol/L, postprandial blood glucose (PPG)>10mmol/L), 10 mg qd of Henagliflozin Proline was sequentially added. If the blood glucose levels did not meet the standard after 4 weeks of treatment (FPG>7mmol/L, PPG>10mmol/L), 100 mg qd of Ruigeliflozin was added
  Interventions: Drug: Sequential treatment group

INTERVENTIONS:
Drug: Combination therapy — Henagliflozin Proline 10 mg qd+Regagliptin 100 mg qd+Metformin 500mg bid. The dose of metformin from the first to second week is 500mg bid, and the dose from the third to fourth week is 1000mg bid. If the maximum dose of metformin cannot be tolerated, the researcher shall increase the dosage according to the patient's tolerance situation. The minimum dose is 1000mg/day.
  Arms: Combination therapy
Drug: Sequential treatment group — Metformin, the dose from the first to second week is 500mg bid, and the dose from the third to fourth week is 1000mg bid. If the maximum dose of metformin cannot be tolerated, the researcher shall increase the dosage according to the patient's tolerance situation. The minimum dose is 1000mg/day. After the fourth week of treatment, blood glucose levels were measured. For those whose blood glucose levels did not meet the standard (fasting blood glucose (FPG)>7mmol/L, postprandial blood glucose (PPG)>10mmol/L), 10 mg qd of Henagliflozin Prolinewas sequentially added. If the blood glucose levels did not meet the standard after 4 weeks of treatment (FPG>7mmol/L, PPG>10mmol/L), 100 mg qd of Ruigeliflozin was added
  Arms: Sequential treatment group

SUMMARY:
This study evaluated the efficacy and safety of initial combined treatment of Henggliptin, Retagliptin and Metformin by including new type 2 diabetes patients. This study is a multicenter, randomized, open label, positive control study. It is planned to include 160 new type 2 diabetes patients who meet the inclusion criteria of the study. The study is divided into three stages: screening period (V0, -14d-0), treatment period (V1-V8, D1-24w) and safe follow-up period (V9, 28w), with a total of 10 planned visits. This study was divided into an experimental group and a control group. The experimental group received a one-time addition of 10 mg qd of Henggliptin, 100 mg qd of Regagliptin, and 500mg of Metformin. The control group was first treated with metformin. If the blood sugar level did not meet the standard (fasting blood glucose (FPG)>7mmol/L, postprandial blood glucose (PPG)>10mmol/L), Henggeliflozin 10 mg qd was sequentially added. If the blood sugar level did not meet the standard after 4 weeks, Regagliptin 100 mg qd was added. During the follow-up period, evaluate blood glucose control, pancreatic islet function, and safety in both groups of patients.

ELIGIBILITY:
Inclusion Criteria:

1. Untreated newly diagnosed T2DM patients;
2. Age ≥ 18 years old;
3. 8.0% ≤ HbA1c<11.0%;
4. 19 kg/m2 ≤ BMI<35 kg/m2;
5. eGFR ≥ 60 ml/min1.73m2;
6. Voluntarily participate and sign an informed consent form

Exclusion Criteria:

1. Pregnant and lactating women, as well as women of childbearing age who are unwilling to take reliable contraceptive measures;
2. Individuals who are known to be allergic to Henggliflozin, Regagliptin, or Metformin;
3. Other types of diabetes except type 2 diabetes;
4. Type 2 diabetes with a history of ketoacidosis (DKA) in the last 6 months;
5. NYHA cardiac grade IV patients;
6. Within 30 days prior to the screening visit, admission due to acute coronary syndrome (ST segment elevation myocardial infarction, non ST segment elevation myocardial infarction, or unstable angina), percutaneous coronary intervention, or cardiac surgery; Or plan to undergo percutaneous coronary intervention or cardiac surgery within 3 months.
7. Confirmed respiratory system diseases (such as chronic obstructive pulmonary disease, pulmonary arterial hypertension, etc.);
8. History of acute or chronic pancreatitis;
9. Uncontrolled hypertension, defined as systolic blood pressure ≥ 160 mmHg and/or diastolic blood pressure ≥ 100 mmHg (average of three supine blood pressure measurements) during screening visits;
10. Patients with orthostatic hypotension and/or systolic blood pressure<90 mmHg at visit 0 or visit 1, or clinically diagnosed as having low blood volume;
11. Diagnosed malignant tumor patients with an expected life expectancy of less than 1 year;
12. Patients with a history of recurrent urinary and reproductive tract infections (judged by clinical doctors);
13. Patients who participate in other clinical trials within 3 months;
14. Alcohol or drug addiction.
15. In addition to the above, the researchers determined that patients who are not suitable to participate in this clinical trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2024-05-31 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of subjects with HbA1c<7% at 12w | From enrollment to the end of treatment at 12 weeks

SECONDARY OUTCOMES:
The proportion of subjects with HbA1c<7% at week 24 | From enrollment to the end of treatment at 24 weeks
The proportion of subjects with HbA1c<6.5% at 12 week | From enrollment to the end of treatment at 12 weeks
The proportion of subjects with HbA1c<6.5% at 24 week | From enrollment to the end of treatment at 24 weeks
Changes in HbA1c compared to baseline at 12 weeks | From enrollment to the end of treatment at 12 weeks
Changes in HbA1c compared to baseline at 24 weeks | From enrollment to the end of treatment at 24 weeks
Changes in fingertip blood glucose (seven point blood glucose spectrum) compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in 2hPPG compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in FBG compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in systolic pressure compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in diastolic pressure compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in body weight compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in waist circumference compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in eGFR compared to baseline at 4w, 8w, 12w, and 24w | From enrollment to the end of treatment at 4/8/12/24 weeks
Changes in C-peptide levels during the 12 and 24 weeks compared to baseline during abdominal and 2-hour postprandial periods | From enrollment to the end of treatment at 12 and 24 weeks
Changes in insulin levels during the 12 and 24 weeks compared to baseline during abdominal and 2-hour postprandial periods | From enrollment to the end of treatment at 12 and 24 weeks

IPD SHARING:
Plan to Share IPD: Undecided